CLINICAL TRIAL: NCT00866099
Title: Evidence-based Interventions In Dementia EVIDEM-ED: Early Recognition and Response in Primary Care
Brief Title: Dementia Early Recognition and Response in Primary Care
Acronym: EVIDEM-ED
Status: Unknown | Phase: Phase 2 / Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: University College, London (Other)
Collaborators: National Institute for Health Research, United Kingdom (Other Government); Central and North West London NHS Foundation Trust (Other); King's College London (Other); University of Hertfordshire (Other); St George's, University of London (Other); London School of Economics and Political Science (Other); Imperial College London (Other)
Responsible Party: Professor Steve Iliffe, University College London
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: FIS No: 49287; Award Code: GZFP
Record Dates: First submitted 2009-03-19; First posted 2009-03-20 (Estimated); Last update posted 2010-04-19 (Estimated); Status verified 2009-03

CONDITIONS: Dementia
Keywords: Dementia; primary care; early diagnosis; psychosocial interventions; cholinesterase inhibitors
MeSH Terms: conditions — Dementia; Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- "Normal Care" (No Intervention): Primary care practices randomly allocated will be given a summary of the NICE/SCIE dementia guidelines (2006) and offered workshop training and software at the end of the study.
- Training (Experimental): Practices randomly allocated to the intervention arm will be asked to participate in tailored learning activities on dementia, over a three-month period and will be given an electronic training manual (based on Microsoft packages) which they can run in the background during and after consultations with people with known or suspected dementia syndrome and face-to- face individualised workshop sessions.
  Interventions: Other: Educational Dementia training

INTERVENTIONS:
Other: Educational Dementia training — Tailored learning activities on dementia, over a three-month period and will be given an electronic training manual (based on Microsoft packages) which they can run in the background during and after consultations with people with known or suspected dementia syndrome and face-to- face individualised workshop sessions.
  Tailoring of the education programme is carried out in a three step process: 1) an educational needs analysis is carried our using a standard checklist to identify aspects of dementia care which the practice perceives as problematic for them; 2) a prescription for education is then written to address shortcomings; 3) the best forms of learning are then identified.
  Arms: Training

SUMMARY:
The purpose of this study is to develop and test an educational intervention for dementia in primary care, combining timely diagnosis, psychosocial support around the period of diagnosis and management concordant with guidelines.

DETAILED DESCRIPTION:
Dementia presents many challenges for primary care. Early diagnosis is important as this allows those with dementia and their family care networks to engage with support services and plan for the future. These actions can relieve the significant psychological distress that people with dementia and close supporters may experience , and provide knowledge about the availability of medical and psycho-social support that can improved functioning and morale

The main efforts to improve the identification and diagnosis of dementia should logically be targeted at primary care as this is the first point of contact for most individuals and their carers when faced with experiences of 'ill health'. There is, however, evidence that dementia remains under-detected and sub-optimally managed in general practice . An educational intervention that could enhance clinical practice, improving the skills of practitioners in the recognition of and response to dementia syndromes, could therefore be beneficial to people with dementia and their families, and potentially to health and social services.

ELIGIBILITY:
Inclusion Criteria:

* Patients with memory or other cognitive impairments suggestive of dementia syndrome
* those with a formal diagnosis of dementia, of any type.

Exclusion Criteria:

* Patients and carers who are already involved in concurrent research
* If the key professional feels that an approach to the person with dementia or their carer would be inappropriate, for example the dementia is very severe, or that an approach may increase distress
* and any other important reason that the key professional may have for why the person with dementia or their carer should not be contacted.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 125 (Estimated)
Dates: Start 2009-07; Primary Completion 2011-05 (Estimated); Study Completion 2012-09 (Estimated)

PRIMARY OUTCOMES:
An increase in the proportion of patients with dementia receiving two dementia reviews per year, from 20% to 50% | twelve month follow up

SECONDARY OUTCOMES:
quality of life, met and unmet need in carers and/or people with dementia | twelve month follow up
documented concordance with intervention recommendations on recording disclosure decisions & consequences | twelve month follow up
documented concordance with screening for depression | twelve month follow up
documented concordance with referral to social services | twelve month follow up
documented concordance with informing people with dementia and their carers about relevant local voluntary organisations | twelve month follow up
documented concordance with provision of legal information | twelve month follow up
documented concordance with shared management of cholinesterase inhibitor medication | twelve month follow up

CONTACTS AND LOCATIONS:
Overall Officials: Jane Wilcock, MA(hons) MSc, Principal Investigator — University College, London
Locations (2):
- United Kingdom (2):
  - Department of Primary Care and Population Health, London, England
  - University College London, London, Greater London

REFERENCES:
- [Derived] Wilcock J, Iliffe S, Griffin M, Jain P, Thune-Boyle I, Lefford F, Rapp D. Tailored educational intervention for primary care to improve the management of dementia: the EVIDEM-ED cluster randomized controlled trial. Trials. 2013 Nov 20;14:397. doi: 10.1186/1745-6215-14-397. PMID 24257429
- [Derived] Iliffe S, Wilcock J, Griffin M, Jain P, Thune-Boyle I, Koch T, Lefford F. Evidence-based interventions in dementia: A pragmatic cluster-randomised trial of an educational intervention to promote earlier recognition and response to dementia in primary care (EVIDEM-ED). Trials. 2010 Feb 10;11:13. doi: 10.1186/1745-6215-11-13. PMID 20146803
- See also: programme website — http://www.evidem.org.uk